CLINICAL TRIAL: NCT01000064
Title: Psychostimulant Treatment of TBI-Related Attention Deficits: fMRI Analysis of Neural Mechanisms of Response
Brief Title: Treatment of Traumatic Brain Injury (TBI)-Related Attention Deficits
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: unable to meet recruitment goals
Sponsor: Vanderbilt University (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Michael G. Tramontana, Associate Professor of Psychiatry, Neurology, and Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TBI 090563
Record Dates: First submitted 2009-10-15; First posted 2009-10-22 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Traumatic Brain Injury; Attention Deficit Disorder
Keywords: Traumatic Brain Injury; Attention Deficit; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vyvanse (Active Comparator): Vyvanse capsule, 30-70 mg, each morning for 6 weeks.
  Placebo capsule each morning for 6 weeks.
  Brain scans (fMRI) performed at baseline, 6th week visit and 12th week visit.
  Interventions: Drug: Vyvanse; Procedure: fMRI; Drug: Placebo
- Placebo (Placebo Comparator): Vyvanse capsule, 30-70 mg, each morning for 6 weeks.
  Placebo capsule each morning for 6 weeks.
  Brain scans (fMRI) performed at baseline, 6th week visit and 12th week visit.
  Interventions: Drug: Vyvanse; Procedure: fMRI; Drug: Placebo

INTERVENTIONS:
Drug: Vyvanse — 30 mg - 70 mg capsules taken every morning for 6 weeks.
Procedure: fMRI — Brain scans (fMRI) performed at baseline, 6 week visit and 12th week visit.
  Other Names: functional magnetic resonance imaging
Drug: Placebo — Placebo capsules taken every morning for 6 weeks.

SUMMARY:
The purpose of this research study is to evaluate whether Vyvanse, a psychostimulant, can help with attention deficits due to traumatic brain injury (TBI). Vyvanse is currently approved for the treatment of Attention-Deficit/Hyperactivity (ADHD). The exact effects this drug may have on attention deficits caused by TBI are not known, but we expect that Vyvanse will be of some help in treating those types of problems as well. The study will utilize functional magnetic resonance imaging (fMRI) methods, as well as neurobehavioral measures, to elucidate neural mechanisms of response.

DETAILED DESCRIPTION:
Symptoms of inattentiveness, impulsivity, and poor persistence have been observed in both children and adults following traumatic brain injury (TBI). These often are among the most prominent symptoms manifested and may contribute to interference in a variety of other functional domains. Although there has been some use of psychostimulant medication to treat TBI-acquired attention deficits, it remains a relatively uncommon clinical practice. This study, by highlighting mechanisms of action, could serve to promote the appropriate use of this type of treatment for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 16 to 45
* Closed head injury rated as moderate/severe (based on Glasgow Coma Scale rating, estimated posttraumatic amnesia, etc.)
* Sustained 6 to 36 months earlier, and considered to be neurologically stable
* Persistent (> 6 months) problems with focused or sustained attention (+1 SD or worse on Inattention component of ADHD self ratings) corroborated by professional staff (nurses, therapists, etc.) or caregivers. Problems with attention/concentration rated as among most prominent cognitive changes.
* Accompanying features may include diminished arousal/speed/stamina and/or disinhibited symptoms

Exclusion Criteria:

* Penetrating head injury
* Pre-injury history of diagnosed ADHD
* Other psychiatric conditions such as mania or psychosis. Current posttraumatic stress disorder (PTSD) symptoms may be present but not so severe as to require pharmacologic treatment.
* Lifetime history of psychostimulant abuse or dependence. Other (non-psychostimulant) substance abuse within the past 6 months. Total lifetime drug use will not exceed 5 times each for substances such as amphetamine, meth-amphetamine, or cocaine.
* Prior treatment with psychostimulant(s)
* Tics or other contraindications for psychostimulant use including arteriosclerosis, cardiovascular disease, uncontrolled hypertension or hyperthyroidism, glaucoma, agitation, use of MAO inhibitor within 6 weeks
* Current treatment with other psychotropic medication(s) within the past 6 weeks
* Estimated IQ < 80
* Sensory and/or motor impairment(s) seriously limiting testing options
* Other neurological conditions including epilepsy, degenerative disorders, brain tumor, or stroke.
* Physical conditions affecting arousal, activity level or stamina, including uncontrolled thyroid dysfunction, anemia, autoimmune or metabolic disorders, untreated moderate/severe sleep apnea, etc.
* Persons for whom MRI scanning is contraindicated, including weight greater than 275 pounds (due to scanner table limitations), severe claustrophobia, implanted electronic medical devices (e.g. pacemaker, cochlear or other inner ear implant, deep brain stimulator), metallic foreign object in eye or rest of the body, history of sheet metal work, aneurysm clips, non-removable metallic piercings, and dental prosthetics.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Tramontana, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 22 cases enrolled, five were lost prior to the baseline assessment (moved, unable to contact, no-showed). Two cases were left on hold. Two cases met safety end-point criteria before group assignment. This left 13 individuals who were assigned to groups.
Groups:
- Vyvanse First, Then Placebo: Drug: Vyvanse 30 mg for 7 days. 50 mg for 7 days. 70 mg for 28 days.
  Procedure/Surgery: fMRI Brain scans (fMRI) performed 3 times.
  Drug: Placebo Capsules taken for 42 days.
- Placebo First, Then Vyvanse: Drug: Placebo Capsules taken for 42 days.
  Procedure/Surgery: fMRI Brain scans (fMRI) performed 3 times.
  Drug: Vyvanse 30 mg for 7 days. 50 mg for 7 days. 70 mg for 28 days.
Period: Overall Study
Arm/Group | Vyvanse First, Then Placebo | Placebo First, Then Vyvanse
Started | 7 | 6
Completed | 6 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Drug: Vyvanse 30 mg for 7 days. 50 mg for 7 days. 70 mg for 28 days.
  Procedure/Surgery: fMRI Brain scans (fMRI) performed 3 times.
  Drug: Placebo Capsules taken for 42 days.
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.85 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition.
  CPT-II Preservations represent responses in which reaction time was less than 100 ms; these responses are assumed to be anticipatory, random, or slow/inattentive (i.e., carried over from the previous response) because it is physiologically impossible to respond accurately in so short a time. Higher T-scores, percentiles, and means indicate worse performance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
ms | 50.23 (6.67) | 59.76 (17.29)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.053, t-test, 2 sided

2. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition.
  CPT-II Hit Reaction Time (RT) Block Change measures inattention and vigilance. Lower values indicate less slowing in RT as the test progressed. High T-scores indicate decreased vigilance over time.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
t-scores | 47.70 (7.47) | 54.21 (7.68)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.052, t-test, 2 sided

3. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using Conners Continuous Performance Task (CPT-II)
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition.
  CPT-II Hit Reaction Time (RT) Inter-Stimulus Interval (ISI) Change assesses the ability to adapt to changing inter-stimulus intervals. Inter-stimulus intervals refers to the amount of time between presentation of stimuli. High t-scores indicate that RT increased as the ISI increased; negative values indicate that RT decreased as the ISI increased.
  Less Hit RT ISI Change indicates less variability in RT depending on the speed of presentation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
t-scores | 58.08 (17.92) | 65.93 (17.61)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

4. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition.
  CPT-II Hit Reaction Time (RT) Standard Error (SE) measures inattention. Consistency of response times is measured by the standard error for responses to targets. Higher values indicate a greater amount of inattention.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
ms | 54.26 (18.21) | 64.04 (15.68)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

5. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using the Wechsler Adult Intelligence Scale -- Fourth Edition (WAIS-IV) Digit Span-Backward Subtest.
Description: Digit Span repeats strings of digits of increasing length said by the examiner in the same (forward) and in reverse (backward) order. It measures working memory and concentration with a range of scaled scores from 1-19, with higher scaled scores indicating better performance when compared to population norms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 11.60 (3.86) | 9.40 (4.40)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

6. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using the Conners Adult ADHD Rating Scale: Long Form (CAARS:L) "Inattention/Memory Problems" Sub-scale.
Description: The CAARS:L is an assessment tool that prompts an observer to provide valuable information about the client. This instrument is helpful when considering a diagnosis of ADHD or related problem. High scores on the "Inattention/Memory Problems" sub-scale may indicate difficulty in concentration, difficulty planning or completing tasks, forgetfulness, absent-mindedness, and/or being disorganized.
  T-scores (M = 50, SD = 10) are used to measure ratings with higher t-scores indicating greater inattention and memory problems. When a t-score is around 60, this indicates greater risk.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
t-scores | 51.25 (13.29) | 56.33 (12.39)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.040, t-test, 2 sided

7. Primary Outcome: Assessment of Various Components of Attention, Related Cognitive Processes and ADHD Symptoms, Using the Behaviour Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Organization of Materials" Sub-scale.
Description: The BRIEF-A is a standardized rating scale developed to observe everyday behaviors associated with specific domains of the executive functions in adults ages 18 to 90 years. The "Organization of Materials" scale measures orderliness of work, living, and storage spaces.
  T-scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning on the BRIEF-A, with higher scores indicating more difficulty in a particular area.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 13 | 13
t-scores | 48.55 (7.95) | 56.00 (12.76)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

8. Secondary Outcome: Evaluation of Which Types of Patients Are Most Likely to Benefit From Treatment
Time Frame: 12 weeks
Population: No data were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: The Study Will Utilize fMRI Methods (as Well as Aforementioned Neurobehavioral Measures) to Elucidate Neural Mechanisms of Response.
Time Frame: 12 weeks
Population: Based on the analysis of neurobehavioral assessment data, complications with screening, and limited sample size, the neural mechanisms of response to Vyvanse vs placebo were not significant enough to be measured and compared by fMRI. There is no data from the fMRI to be reported because it was abandoned as an aspect of this study before analysis.
Arm/Group | Vyvanse First, Then Placebo | Placebo First, Then Vyvanse
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 14 weeks.
Description: Once enrolled, all cases underwent weekly clinical monitoring, drug trial implementation, as well as safety and compliance assessments by a research nurse at the Vanderbilt Clinical Trials Centre (CTC).
Groups:
- Vyvanse: Drug: Vyvanse 30 mg for 7 days. 50 mg for 7 days. 70 mg for 28 days.
- Placebo: Placebo capsule Taken for 42 days.
Arm/Group | Vyvanse | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Participant withdrawal during study leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No